CLINICAL TRIAL: NCT05365061
Title: Periosteal Electrical Dry Needling With no Maintenance Treatments vs. Maintenance Treatments Every Other Month vs. Maintenance Treatments Once Per Month for Knee Osteoarthritis
Brief Title: Periosteal Electrical Dry Needling for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, Principal Investigator, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT20231
Record Dates: First submitted 2022-04-13; First posted 2022-05-09 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Periosteal electrical dry needling followed by no maintenance treatments (Experimental): Periosteal electrical dry needling followed by no maintenance treatments
  Interventions: Other: periosteal electrical dry needling with no maintenance treatments
- Periosteal electrical dry needling followed by maintenance treatments every other month (Active Comparator): Periosteal electrical dry needling followed by maintenance treatments every other month
  Interventions: Other: periosteal electrical dry needling with maintenance treatments every other month
- Periosteal electrical dry needling followed by monthly maintenance treatments (Active Comparator): Periosteal electrical dry needling followed by monthly maintenance treatments
  Interventions: Other: periosteal electrical dry needling with monthly maintenance treatments

INTERVENTIONS:
Other: periosteal electrical dry needling with no maintenance treatments — periosteal electrical dry needling
  Arms: Periosteal electrical dry needling followed by no maintenance treatments
Other: periosteal electrical dry needling with maintenance treatments every other month — periosteal electrical dry needling with maintenance treatments every other month
  Arms: Periosteal electrical dry needling followed by maintenance treatments every other month
Other: periosteal electrical dry needling with monthly maintenance treatments — periosteal electrical dry needling with monthly maintenance treatments
  Arms: Periosteal electrical dry needling followed by monthly maintenance treatments

SUMMARY:
The purpose of this research is to treat patients with knee osteoarthritis (OA) with periosteal electric dry needling (PEDN). It is also to determine the optimal "maintenance" regiment (i.e. maintenance treatments, one maintenance treatment every other month, or one maintenance treatment per month) required to maintain improvements in pain and function following PEDN. Physical therapists commonly use PEDN to treat knee OA, and previous studies suggest that this treatment is useful for reducing pain and improving function in patients with osteoarthritis. However, an appropriate maintenance treatment strategy to maintain these outcomes is presently unknown.

DETAILED DESCRIPTION:
Patients with knee osteoarthritis will be randomized to receive periosteal electrical dry needling 1-2 treatments per week for 6 weeks (up to 10 sessions total) followed by either: 1. no maintenance treatments, 2. one maintenance treatment every other month or 3. one maintenance treatment per month.

ELIGIBILITY:
Inclusion Criteria:

1. Adult over the age of 18 years old:
2. Report of knee pain of at least 2/10 per NPRS (0---10 scale) for >3 months
3. Report of at least 3 of the following per Altman et al. (1986) (sensitivity = 95% / specificity = 69%)

   1. Over 50 Years of age
   2. Less than 30 minutes of morning stiffness
   3. Crepitus on active motion
   4. Bony tenderness
   5. Bony enlargement
   6. No palpable warmth of Synovium

Exclusion Criteria:

1. Report of red flags to manual physical therapy to include: hypertension, infection, diabetes, peripheral neuropathy, heart disease, stroke, chronic ischemia, edema, severe varicosities, tumor, metabolic disease, prolonged steroid use, fracture, RA, osteoporosis, severe vascular disease, malignancy, etc.
2. History of physical therapy, massage therapy, chiropractic treatment, or injections for knee pain in last 4 weeks.
3. History of a partial or total knee replacement on the painful lower extremity.
4. History of a surgical procedure on either lower extremity in last 12 months.
5. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

   1. Weakness involving a major muscle group of the lower extremity.
   2. Diminished patella or achilles tendon reflex
   3. Diminished or absent sensation to pinprick in lower extremity dermatome.
6. Involvement in litigation or worker's compensation regarding knee pain.
7. Any condition that might contraindicate the use of periosteal electric dry needling
8. The patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC Knee Osteoarthritis Index (Total Score) | baseline, 6 weeks, 14 weeks, 22 weeks, 30 weeks
  24 questions each worth 0-4 points with maximum score of 96 points possible. The greater the score, the worse the symptoms of knee OA

SECONDARY OUTCOMES:
Change in WOMAC Knee Osteoarthritis Index (Pain) | baseline, 6 weeks, 14 weeks, 22 weeks, 30 weeks
  5 questions each worth 0-4 points with maximum score of 20 points possible. The greater the score, the worse the pain.
Change in WOMAC Knee Osteoarthritis Index (Stiffness) | baseline, 6 weeks, 14 weeks, 22 weeks, 30 weeks
  2 questions each worth 0-4 points with maximum score of 8 points possible. The greater the score, the worse the stiffness.
Change in WOMAC Knee Osteoarthritis Index (Physical Function) | baseline, 6 weeks, 14 weeks, 22 weeks, 30 weeks
  17 questions each worth 0-4 points with maximum score of 68 points possible. The greater the score, the worse the physical function.
Change in knee pain | baseline, 6 weeks, 14 weeks, 22 weeks, 30 weeks
  Average Numeric Pain Rating Score. Higher score means greater pain
Change in GROC (Global Rating of Change score) | 6 weeks, 14 weeks, 22 weeks, 30 weeks
  GROC (ranges from -7 to +7). Global Rating of Change score
Change in Medication Intake (Frequency of medication intake during last time period) | baseline, 30 weeks
  Frequency of medication intake during last time period

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, PhD DPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Team Rehabilitation, Chamblee, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dunning J, Young I, Taylor N, Mourad F, Bliton P, Butts R, Escaloni J, Gorby P, Varghese R, Maselli F, Fernandez-de-Las-Penas C. Effect of dose interval of periosteal and intraarticular electrical dry needling boosters on pain and disability in patients with knee osteoarthritis: a multi-center randomized clinical trial. Physiother Theory Pract. 2025 Oct 17:1-14. doi: 10.1080/09593985.2025.2575837. Online ahead of print. PMID 41104706